CLINICAL TRIAL: NCT03498235
Title: Randomized,Double-Blind Trial A Comparative Analysis of the Effects of Sevoflurane and Propofol on Optic Nerve Sheath Diameter During Steep Trendelenburg Position and Pneumoperitoneum for Laparoscopic Gynecologic Surgery
Brief Title: Effects of Sevoflurane and Propofol on Optic Nerve Sheath Diameter During Laparoscopic Gynecologic Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Weilian Geng, Director,Clinical Research, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: V2018-2
Record Dates: First submitted 2018-03-08; First posted 2018-04-13 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Laparoscopic Gynecologic Surgery
Keywords: sevoflurane; propofol; intracranial pressure; optic nerve sheath diameter
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team Sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane
- Team Propofol (Experimental)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — In Team Sevoflurane,patients undergo sevoflurane.
  Arms: Team Sevoflurane
Drug: Propofol — In Team Propofol ,anesthesia is maintained with propofol
  Arms: Team Propofol

SUMMARY:
Intracranial pressure（ICP) increases during laparoscopic gynecologic surgery increase (ICP) and may alter optic nerve sheath diameter(ONSD).This study measures ONSD in different team because sevoflurane and propofol have different effects on ICP.Half of participants will receive sevoflurane anesthesia,while the other half undergo propofol anesthesia.

DETAILED DESCRIPTION:
Due to the anatomical and physiological characteristics of optic nerve sheath ,ONSD increases when ICP rises.

Sevoflurane and propofol have different effects on ICP.When sevoflurane concentration >1.1 minimum alveolar concentration（MAC),ICP increases because of cerebral vasodilatation；on the other hand ,propofol constricts the blood vessels and ICP decreases.

ICP increases during laparoscopic gynecologic surgery because of steep Trendelenburg position and pneumoperitoneum .

Meanwhile,sevoflurane affects self regulation of cerebral blood flow on the way of dose dependent,but propofol has no effects on self regulation of cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status diagnosed as I or II

Exclusion Criteria:

* neuromuscular diseases;laboratory abnormalities in electrolytes; liver and kidney dysfunction;allergy to general anesthetics;pregnancy;ocular lesions including ocular trauma, optic neuritis, optic nerve tumor.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Changes of ultrasonographic optic nerve sheath diameter | from the time when patients enter into operation room to the time when the surgery ending
  different time including pre-anesthesia, after intubation,every 15 minutes in the first hour after beginning of surgery, every hour when one hour after surgery beginning,surgery ending.

SECONDARY OUTCOMES:
Analyzed whether mean arterial pressure influence the change of ONSD based on 110 patients in two groups. | from the time when patients enter into operation room to the time when the surgery ending
  Mean arterial pressure was collected when measures ONSD by ultrasound.
Analyzed whether airway pressure influence the change of ONSD based on 110 patients in two groups. | from the time when patients enter into operation room to the time when the surgery ending
  airway pressure was collected when measures ONSD by ultrasound.
Analyzed whether urine volume influence the change of ONSD based on 110 patients in two groups. | from the time when patients enter into operation room to the time when the surgery ending
  Recording urine volume when the surgery finished.
Analyzed whether blood loss influence the change of ONSD based on 110 patients in two groups. | from the time when patients enter into operation room to the time when the surgery ending
  Recording blood loss when the surgery finished.
Analyzed whether fluid volume influence the change of ONSD based on 110 patients in two groups. | from the time when patients enter into operation room to the time when the surgery ending
  Recording fluid volume when the surgery finished.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geng W, Chen C, Sun X, Huang S. Effects of sevoflurane and propofol on the optic nerve sheath diameter in patients undergoing laparoscopic gynecological surgery: a randomized controlled clinical studies. BMC Anesthesiol. 2021 Jan 27;21(1):30. doi: 10.1186/s12871-021-01243-7. PMID 33504329